CLINICAL TRIAL: NCT00033319
Title: UKCAP Trial: A Multi-Center Double Blind Randomised Controlled Trial Of Aspirin And/Or Folate Supplementation For the Prevention Of Recurrent Colorectal Adenomas
Brief Title: Aspirin and/or Folic Acid in Preventing Recurrent Colorectal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen's Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000069273; QMC-UKCAP; EU-20045
Record Dates: First submitted 2002-04-09; First posted 2003-07-01 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2002-12

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folic Acid; Aspirin

INTERVENTIONS:
Dietary Supplement: folic acid
Drug: acetylsalicylic acid

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of aspirin and/or folic acid may be effective in preventing recurrent polyps in patients who have had polyps removed previously.

PURPOSE: Randomized clinical trial to determine the effectiveness of aspirin and/or folic acid in preventing the recurrence of colorectal polyps.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether aspirin and/or folic acid prevents recurrence of colorectal adenomas in patients who have had colorectal adenomas removed.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral aspirin and oral folic acid daily.
* Arm II: Patients receive oral aspirin and oral placebo daily.
* Arm III: Patients receive oral placebo and oral folic acid daily.
* Arm IV: Patients receive 2 oral placebos daily. In all arms, treatment continues for 3 years in the absence of unacceptable toxicity.

After completion of the 3-year intervention, all patients undergo a surveillance colonoscopy.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 1,300 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenoma removed within the past 6 months

  * Greater than 0.5 cm after fixation or greater than 0.7 cm at time of removal

    * OR
  * Any size with a history of prior colorectal adenoma removal(s)
* Removed via colonoscopy, flexi-sigmoidoscopy (provided barium enema has been performed), or transanal endoscopic microsurgery
* Removal must be considered complete with follow-up to be done within 6 months
* No prior resection of large bowel (e.g., hemi-colectomy or greater, anterior resection, or subtotal colectomy)

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* No active bleeding disorders

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No unstable heart conditions

Pulmonary:

* No unstable asthma

Other:

* Not pregnant and no potential to become pregnant within the next 3 years
* No unstable diabetes
* No active upper gastrointestinal ulceration
* No known aspirin intolerance or sensitivity
* No other serious medical conditions that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No other concurrent folic acid
* No concurrent anticoagulants
* No other prior or concurrent non-steroidal anti-inflammatory drugs, prescribed or self-medicated (more than 3 tablets per week)

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-05

CONTACTS AND LOCATIONS:
Overall Officials: Richard Logan, MD, Study Chair — Queen's Medical Center
Locations (32):
- United Kingdom (32):
  - Antrim Hospital, Antrim, England
  - City Hospital - Birmingham, Birmingham, England
  - Birmingham Heartlands and Solihull NHS Trust (Teaching), Birmingham, England
  - Southmead Hospital, Bristol, England
  - Frenchay Hospital, Bristol, England
  - Bristol Royal Infirmary, Bristol, England
  - Derby City General Hospital, Derby, England
  - Wordsley Hospital, Dudley, England
  - Glenfield Hospital, Leicester, England
  - Royal Liverpool and Broadgreen Hospitals, Liverpool, England
  - Manchester Royal Infirmary, Manchester, England
  - Wythenshawe Hospital, Manchester, England
  - Trafford General Hospital, Manchester, England
  - Southport and Formby District General Hospital, Merseyside, England
  - Merthyr Tydfil Hospital, Merthyr, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Queen's Medical Centre, Nottingham, England
  - Whiston Hospital, Prescot Merseyside, England
  - Salford Royal Hospitals NHS Trust, Salford, England
  - Sheffield Teaching Hospitals, Sheffield, England
  - Northern General Hospital, Sheffield, England
  - Solihull Hospital, Solihull, England
  - Royal Victoria Hospital, Belfast, Northern Ireland
  - Whiteabbey Hospital, Newtownabbey, Northern Ireland
  - Princess of Wales Hospital, Bridgend, Wales
  - University of Wales College of Medicine, Cardiff, Wales
  - Selly Oak Hospital, Birmingham
  - East Glamorgan Hospital, Lhantrisant
  - North Manchester Healthcare NHS Trust, Manchester
  - Royal Gwent Hospital, Newport Gwent
  - King's Mills Hospital, Nottinghamshire
  - Rotherham District General Hospital-NHS Trust, Rotherham